CLINICAL TRIAL: NCT04811404
Title: A PET Study With [11C]PBR-28 and an Experimental Medication, Ethyl Eicosapentaenoic Acid
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Reassessment of rationale for study
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Martin Lan, Assistant Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8044
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — eicosapentaenoic acid ethyl ester; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ethyl eicosapentaenoic acid (Experimental): Ethyl eicosapentaenoic acid will be given at 1G by mouth twice per day
  Interventions: Drug: Ethyl Eicosapentaenoic Acid

INTERVENTIONS:
Drug: Ethyl Eicosapentaenoic Acid — Treatment will be for six weeks
  Other Names: Ethyl EPA; icosapent ethyl

SUMMARY:
This pilot study will ask whether omega three fatty acids have an antidepressant effect in bipolar depression by decreasing brain inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Diagnosis of of bipolar I or bipolar 2 disorder and currently meets criteria for a major depressive episode
3. Depression of sufficient severity to score at least 16 on the first 17 items of the Hamilton Depression Rating Scale including the atypical depression items addendum at the time of recruitment
4. Age range 18-60
5. Females of child-bearing potential must be willing to use an acceptable method of birth control throughout the study. These include abstinence, birth control pill, male condom, IUD, depo-provera, Norplant male sterilization, female sterilization
6. Not taking more than two psychotropic medications at time of recruitment to avoid polypharmacy. Participants will not have changed the dose of the medication for at least 8 weeks before enrollment.

   Only participants with bipolar 2 disorder diagnosis may be off psychotropic medications at time of enrollment. In that case, they must not have stopped any medications within 8 weeks of enrollment.

   Participants can be taking diphenhydramine but no benzodiazepines or other hypnotics as needed at time of enrollment.
7. Genotyping as a medium or high TSPO binding type

Exclusion Criteria:

1. Diagnosis of any other major psychiatric disorders such as lifetime schizophrenia, schizoaffective disorder, current psychotic features of bipolar disorder, or recent moderate substance use disorder (within 4 months of recruitment); IV drug use. Meets DSMV criteria for a manic episode, or Young Mania Rating Scale score >12, at the time of screening.
2. Previous failed trial or intolerable side effects of ethyl EPA or any other form of omega 3 fatty acids
3. A first-degree family history of schizophrenia if the participant is less than 33 years old.
4. Significant active physical illness, including blood dyscrasias, lymphomas, hypersplenism, endocrinopathies, renal failure, chronic obstructive lung disease, autonomic neuropathies, peripheral vascular disease. Any disorders with inflammation, malignancy, autoimmune or infectious etiology. Systemic blood pressure >140 or diastolic blood pressure >100. Hemoglobin <11 in females or <13 in males.
5. Actively suicidal, as defined by expressing ideation with a plan or intent for suicide or develops suicidal ideation that requires immediate medical or treatment intervention.
6. Pregnancy, abortion or miscarriage in the two months prior to enrollment or plans to conceive during the course of the study participation
7. Lactating Women
8. ECT within the last 6 months
9. Participants who endorse a history of prior head trauma and score 1.5 standard deviations below the mean on Trailmaking A & B test
10. Metal implants, pacemaker, metal prostheses, metal orthodontic appliances or shrapnel in the body
11. Current, past or anticipated exposure to radiation, including

    1. Having been badged for radiation exposure in the workplace
    2. Participation in nuclear medicine protocols in the last year* *Participants will be eligible, however, if the injected dose and dosimetry of the radiotracer are known and the cumulative annual exposure of the previous studies and this study is lower than the annual limit for research participants defined by FDA (21 CFR 361.1)
12. History of claustrophobia that would prevent the participation in neuroimaging
13. Weight >350 lbs or inability to fit into the MRI scanner**

    ** If there are doubts that the MRI scanner can accommodate the physical dimensions of the participant, the participant's circumference may be measured to determine if it is less than the MR scanner limit of 55 cm. The participant may also be brought to the MRI Center and the MRI technologist will assess whether the participant will be able to fit into the MRI scanner. Metal screening and urine pregnancy testing will be done in this circumstance before the participant enters the MRI area.
14. Current anticoagulant or anti-platelet treatment including aspirin if needed daily
15. Risks of delay to treatment of known efficacy (up to 9 weeks) are too great for the participant. Risks to consider include A) Severity of presenting symptoms B) History of symptom fluctuations or deterioration C) Psychosocial conditions that make delay to treatment unreasonable

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Rating Scale | Six weeks
  Minimum value of 0, maximum value of 60; Greater score reflects greater depression severity

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute/Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No